CLINICAL TRIAL: NCT04917367
Title: Second Affiliated Hospital, College of Medicine, Zhejiang University
Brief Title: Diagnosis and Treatment of Foreign Bodies Outside Pharynx and Esophagus Lumen
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-152
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2021-06

CONDITIONS: Surgery
Keywords: Migrating foreign body; Upper aerodigestive tract; Neck; Laryngoscopy endoscopy; Positioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional surgery group: Conventional surgery with Preoperative foreign body localization
  Interventions: Procedure: exploratory surgery
- New surgery group: new surgery with Intraoperative localization of foreign body
  Interventions: Procedure: exploratory surgery

INTERVENTIONS:
Procedure: exploratory surgery — For foreign bodies in the retropharyngeal space or parapharyngeal space above the esophageal entrance, close to the laryngopharynx cavity with large operating space, suspension laryngoscopy is the first choice according to the principle of proximity. In all cases, a lateral cleft laryngoscope was used to expose the posterior or lateral wall of the laryngopharynx, and 30° endoscope or microscope was used according to the skills of the surgeon.
  For a foreign body below the esophageal entrance, the lateral cervical incision was the first choice due to the small operating space of oral exposure. The lateral cervical incision and other open surgical methods are used for foreign bodies below the entrance of the esophagus or in the submaxillary space or for the anterior cervical band muscle foreign bodies.
  Other Names: lateral cervical incision surgery

SUMMARY:
Objective: To improve the success rate of the treatment of migrating foreign bodies in the upper aerodigestive tract.

Methods: The medical records of inpatients conforming to the diagnosis of migrating foreign bodies between 2020 and 2025 were reviewed. Data regarding age, gender, time from onset to hospitalization, computed tomography (CT) and endoscopic scans, surgical procedures，and follow-up were collected.

ELIGIBILITY:
Inclusion Criteria:

* The foreign body of pharynx or esophagus was confirmed by surgical exploration

Exclusion Criteria:

* The foreign body is in the pharynx or esophagus or is not found during surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People from vulnerable groups are excluded
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate | 5 years
  Success rate of two groups

SECONDARY OUTCOMES:
surgery time | intraoperative
  Surgery time of two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Gang Duan, doctor, Study Director — Second Affiliated Hospital, College of Medicine, Zhejiang University
Locations (1):
- Department of Otolaryngology, Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided